CLINICAL TRIAL: NCT06083597
Title: Development of a Patient-reported Outcome (PRO) Measure for Women With Chronic Pelvic Pain (CPP)
Brief Title: Development of a Patient-reported Outcome Measure for Women With Chronic Pelvic Pain
Acronym: PROM for CPP
Status: Enrolling by invitation | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Society of Interventional Radiology Foundation (Other); Evidera (Industry)
Responsible Party: Sponsor
Other Study IDs: 23-02025699
Record Dates: First submitted 2023-08-31; First posted 2023-10-16 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pelvic Pain Syndrome; Pelvic Congestive Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic pelvic pain of venous origin: Women who are thought to have chronic pelvic pain of venous origin will be interviewed to determine the impacts of their pain on physical, social and emotional aspects of their health and well being.
  Interventions: Other: Qualitative interview
- Chronic pelvic pain of non-venous origin: Women who are thought to have chronic pelvic pain of a non-venous origin will be interviewed to determine the impacts of their pain on physical, social and emotional aspects of their health and well being. They will be asked of the concepts identified by the women with venous origin CPP apply to them and if the impacts of the pain are similar or differ.
  Interventions: Other: Qualitative interview

INTERVENTIONS:
Other: Qualitative interview — Qualitative interviews will be performed on women with chronic pelvic pain of venous origin.

SUMMARY:
The purpose of this study is to develop a patient questionnaire that can be utilized to assess the benefit of treatments of chronic pelvic pain in research studies.

The information collected from a series of patient interviews will lead to the development of a questionnaire that accounts for the full impact of chronic pelvic pain from an affected woman's perspective.

DETAILED DESCRIPTION:
The purpose of this study is to develop a patient-reported outcome (PRO) instrument that can be utilized as an efficacy endpoint to assess medical and surgical treatments of chronic pelvic pain (CPP) in comparative outcomes research.

This instrument will be developed consistent with Food and Drug Administration (FDA) guidance to be appropriate as an efficacy measurement in a clinical trial. The development of such a PRO measure is iterative, and this research protocol includes the qualitative research to develop a draft measure and document content validity. Content validity is first assessed through concept elicitation interviews, followed by cognitive interviews.

Patients who are eligible and consent to participate will:

1. complete a series of standardized health questionnaires
2. participate in an interview with a scientist who is an expert at developing this kind of PRO instrument who will ask patients about the impacts of their COO on their overall health and well being.

The information collected from a series of these interviews will lead to the development of a draft questionnaire which will then be reviewed with additional women with similar causes of CPP as well as with women with other causes of CPP to determine its usability and accuracy at assessing the impacts of CPP on their health and well being.

A final version of the PROM instrument will then be shared with women with CPP before and after any treatment to determine its ability to identify changes in their health and wellbeing.

ELIGIBILITY:
I. First phase of study evaluation women with presumed venous origin chronic pelvic pain

Inclusion Criteria :

1. Non-menopausal women ≥18 years old.

   a. Women who are not menstruating because of ovarian suppression therapy for CPP are eligible.
2. CPP meeting the American College of Obstetricians and Gynecologists criteria.
3. Patient pain is primarily of pelvic and/or pelvic floor origin. Patient may experience other pain symptoms, including bowel, bladder, musculoskeletal, skin allodynia and hyperalgesia, or lower extremity venous or vulvar pain.
4. Imaging demonstrating multiple tortuous pelvic varicose veins > 5 mm in diameter in the ovarian, utero vaginal, and/or uterine arcuate venous plexus.

   a. Imaging must be documented from trans vaginal ultrasound, trans abdominal ultrasound, magnetic resonance imaging, computed tomography, catheter venogram, or trans fundal pelvic venogram. If laparoscopic images are available to confirm veins this size, this would be acceptable as well.
5. Venous contribution to CPP, as determined by clinical impression from a CPP specialist. Clinical impression will be based on the presence of the following symptoms and physical findings:

   a. Symptoms: i. CPP increased with standing, walking, or lifting ii. CPP increased at the end of the day iii. CPP improved by laying down iv. Sexually provoked prolonged post-coital ache b. Physical findings: i. Adnexal tenderness on gentle bimanual exam ii. Tenderness at the ovarian point trans-abdominally iii. Tenderness of the uterus
6. Participant can read, communicate clearly, and understand English or Spanish.
7. Participant is willing and able to participate in an interview and complete questionnaires.
8. Participant is willing and able to provide informed consent.

Exclusion Criteria:

1. Pain symptoms should primarily be of pelvic and/or pelvic floor origin (inclusion criteria #3 above). Pain should not be exclusively low back, hips, symphysis, allodynia or hyperalgesia of the skin, or from varicose veins of the vulvar and/or lower extremities.
2. Pain thought primarily to be due to endometriosis, pelvic floor myalgia, a musculoskeletal etiology, irritable bowel disease, or painful bladder syndrome/interstitial cystitis.
3. Obvious endometriosis based on physical exam or laparoscopy findings.
4. Patients previously treated with a technically successful surgery or vascular procedure for a venous disorder of the pelvis or renal vein.
5. Participant has any clinically relevant medical condition (e.g., severe co morbid condition, severe mental illness, severe visual or auditory impairment, or cognitive impairment) that, in the opinion of the investigator, would interfere with participating in an interview and/or completing the study procedures

II. Second phase of study evaluation women with non-venous origin chronic pelvic pain

Inclusion Criteria :

1. Non-menopausal women ≥18 years old.

   a. Women who are not menstruating because of ovarian suppression therapy for CPP are eligible.
2. CPP meeting the American College of Obstetricians and Gynecologists criteria.
3. Patient pain is primarily of pelvic and/or pelvic floor origin. Patient may experience other pain symptoms, including bowel, bladder, musculoskeletal, skin allodynia and hyperalgesia, or lower extremity venous or vulvar pain.
4. Imaging demonstrating multiple tortuous pelvic varicose veins > 5 mm in diameter in the ovarian, utero vaginal, and/or uterine arcuate venous plexus.

   a. Imaging must be documented from trans vaginal ultrasound, trans abdominal ultrasound, magnetic resonance imaging, computed tomography, catheter venogram, or trans fundal pelvic venogram. If laparoscopic images are available to confirm veins this size, this would be acceptable as well.
5. Venous contribution to CPP, as determined by clinical impression from a CPP specialist. Clinical impression will be based on the presence of the following symptoms and physical findings:

   a. Symptoms: i. CPP increased with standing, walking, or lifting ii. CPP increased at the end of the day iii. CPP improved by laying down iv. Sexually provoked prolonged post-coital ache b. Physical findings: i. Adnexal tenderness on gentle bimanual exam ii. Tenderness at the ovarian point trans-abdominally iii. Tenderness of the uterus
6. Participant can read, communicate clearly, and understand English or Spanish.
7. Participant is willing and able to participate in an interview and complete questionnaires.
8. Participant is willing and able to provide informed consent.

Exclusion Criteria:

1. Pain symptoms should primarily be of pelvic and/or pelvic floor origin (inclusion criteria #3 above). Pain should not be exclusively low back, hips, symphysis, allodynia or hyperalgesia of the skin, or from varicose veins of the vulvar and/or lower extremities.
2. Pain thought primarily to be due to endometriosis, pelvic floor myalgia, a musculoskeletal etiology, irritable bowel disease, or painful bladder syndrome/interstitial cystitis.
3. Obvious endometriosis based on physical exam or laparoscopy findings.
4. Patients previously treated with a technically successful surgery or vascular procedure for a venous disorder of the pelvis or renal vein.
5. Participant has any clinically relevant medical condition (e.g., severe co morbid condition, severe mental illness, severe visual or auditory impairment, or cognitive impairment) that, in the opinion of the investigator, would interfere with participating in an interview and/or completing the study procedures

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Menstruating women
Study Population: Women with chronic pelvic pain (CPP) meeting the American College of Obstetricians and Gynecologists criteria.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1 qualitative concept elicitation interview | 1 month
  Phase 1 qualitative interview about VO-CPP (Chronic pelvic pain originating from venous contribution) signs, symptoms, and impacts, from which a novel VO-CPP questionnaire (PeVD HRQoL) will be drafted, and ultimately assessed for content validity in the Phase 2 interviews. This Phase 1 interview will be conducted with subjects with VO-CPP.

SECONDARY OUTCOMES:
Phase 2 Qualitative cognitive interview | 1 month
  Phase 2 qualitative interview will include questions about item clarity, how the participants interpret the items, ease of completing the PeVD HRQoL questions, questionnaire comprehensiveness, and the appropriateness of the questionnaire format and response scales. This Phase 2 interview will be conducted with subjects with VO-CPP.
Phase 2 qualitative open-ended concept elicitation questions | 1 month
  Phase 2 qualitative open-ended concept elicitation questions. This Phase 2 interview will be conducted with subjects with chronic pelvic pain originating from non-venous causes (NVO-CCP).
Phase 2 qualitative cognitive interview | 1 month
  Phase 2 qualitative interview about the content validity of the novel questionnaire, PeVD HRQoL, with subjects with chronic pelvic pain originating from non-venous causes (NVO-CCP).

CONTACTS AND LOCATIONS:
Overall Officials: Neil M Khilnani, MD, Principal Investigator — Weill Medical College of Cornell University; Robin Pokrzywinski, PhD, Study Director — Evidera
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, informed consent forms, de-identified data, analytic process and the clinical study report will be available for other researchers. The final patient reported outcome instrument will be made available for use by any investigator for clinical research by the study funder SIR Foundation
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anticipated January 2025
Access Criteria: The study protocol, consents and data supporting the PROM instrument will be made available for research purposes to investigators by the study PI. The final patient reported outcome instrument will be made available for use by any investigator for clinical research by license by the study funder SIR Foundation